CLINICAL TRIAL: NCT06451419
Title: Prospective and Controlled Glucocerebrosidase-related Parkinson's Disease Evaluation of Non Motor Symptoms (PROGENS-PD)
Brief Title: Non Motor Symptoms in Glucocerebrosidase-related Parkinson's Disease
Acronym: PROGENS-PD
Status: Enrolling by invitation | Type: Observational
Sponsor: Juan Pablo Romero. MD, PhD (Other)
Collaborators: Fundación de Investigación Biomédica - Hospital Universitario de La Princesa (Other)
Responsible Party: Sponsor-Investigator, Juan Pablo Romero. MD, PhD, Clinical professor, Universidad Francisco de Vitoria
Organization: Universidad Francisco de Vitoria (Other)
Other Study IDs: 5564
Record Dates: First submitted 2024-05-21; First posted 2024-06-11 (Actual); Last update posted 2024-06-28 (Actual); Status verified 2024-06

CONDITIONS: Parkinson Disease
Keywords: glucocerebrosidase heterozygous mutation; non motor symptoms; neuropsychology; posturography
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Glucocerebrosidase associated Parkinson's disease: Patients aged under 70 when symptoms began or with family history of Parkinson's disease who underwent a genetic testing including a pannel of 64 genes associated with Parkinson's diasease and who tested positive for heterozygous glucocerebrosidase mutation.
  Interventions: Other: Tests on non motor symptoms
- Non glucocerebrosidase associated Parkinson's diasease: Patients aged under 70 when symptoms began or with family history of Parkinson's disease who underwent a genetic testing including a pannel of 64 genes associated with Parkinson's diasease and who tested negative for all the mutations in the pannel.
  Interventions: Other: Tests on non motor symptoms

INTERVENTIONS:
Other: Tests on non motor symptoms — Neurological, neuropsychological and self-administered tests on non motor symptoms, including posturography and speed reaction times.

SUMMARY:
The goal of this observational study is to describe non motor symptoms in a prospective study of patients with Parkinson's disease associated to glucocerebrosidase (GBA-PD) mutations.

The main questions it aims to answer are:

* Do GBA-PD patients have a greater burden of non motor symptoms?
* How do these non motor symptoms evolve during a prospective follow up of two years?
* Are these non motor symptoms different from those that affect Parkinson's disease patients without glucocerebrosidase mutations (non GBA-PD), in prevalence, severity and type?
* Do these non motor symptoms correlate with objective measures such as posturography or speed reaction tests?
* Is there a test or combination of tests that can predict the appearance of early or severe non motor symptoms?

For this reason researchers will compare the GBA-PD group of patients with a group of non mutated GBA Parkinson disease.

Participants will undergo a neurological and neuropsychological evaluation with different tests in subsequent visits for a total of 2 years.

DETAILED DESCRIPTION:
Parkinson's disease is the second most prevalent neurodegenerative disorder worldwide. Up to date, the main risk factor for its development is carrying an heterozygous mutation in glucocerebrosidase gene (GBA). GBA codifies for a GC-ase protein that takes part in lysosomal function. The homozygous mutation of this gene gives rise to Gaucher disease, which is a lysosomal disorder. This gene has also been associated with Lewy body dementia.

The presence of an heterozygous mutation in GBA in Parkinson's disease can be found in up to 5-15% of the patients, depending on age and ethnicity. It has been described that those patients carrying the mutation can have an earlier debut of the disease.

According to non motor symptoms, patients are prone to develop earlier and more severe motor symptoms. This has been studied specially in cognitive impairment but also dysautonomia, impulse control disorder and others.

In relation to cognitive impairment these patients usually develop an earlier and more severe affection, reaching dementia states earlier in the disease. Some studies have described a worsening in cognitive function in GBA mutated patients after deep brain stimulation (DBS) to treat parkinsonian symptoms. This prevents patients from being candidates to therapies such as DBS.

For this reason, the investigators consider it important to make a proper description of non motor symptoms in GBA mutated parkinsonian patients, since this finding can help to delineate the prognosis and choose individualized treatments, regarding the suggested differences with other Parkinson's disease patients.

It is an observational prospective cohort study. Participants will be collected from a subgroup of patients that have agreed to undertake a genetic test including a panel of genes associated to Parkinson's disease.

According to the results, patients will be subdivided in two groups according to their genetic status:

* GBA heterozygous mutations
* Absence of genetic mutations

These patients will undergo neurologic evaluations, neuropsychological evaluations and self-administered evaluations. There will be no intervention.

The pharmacologic and other type of treatment assessments will be conducted during their regular follow up with their neurologist.

These visits will be repeated every 6 months for a total of 2 years. Total of 5 visits for each patient.

ELIGIBILITY:
Inclusion Criteria:

* Aged over 18 years old.
* Fulfill Parkinson's disease criteria of Movement Disorder Society 2015.
* Parkinson's disease symptoms began before they were 70 and/or Parkinson's disease family history.
* Underwent a genetic test of Parkinson's disease related genes.
* Heterozygous mutation of glucocerebrosidase gene (only cases).
* Absence of mutation in the Parkinson's disease genetic test (only controls).

Exclusion Criteria:

* Suspicion of atypical parkinsonism.
* Personal history of other neurodegenerative disorders such as Alzheimer's disease.
* Personal history of significant cerebrovascular damage, intracraneal lessions or important craneoencephalic trauma.
* Deep brain stimulation treatment for Parkinson's disease.
* Moderate or severe dementia that precludes from performing the tests.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Parkinson's disease patients whose symptoms began before they were 70 and/or those who had Parkinson's disease family history and underwent a genetic test including the following Parkinson's disease related genes: ADCY5, ANO, APOE, APP, ATP1A3, ATP9A, C19orf12, CHCHD2, CNEP1R1, COX20, CTDNEP1, DCTN1, DNAJC13, DNAJC6, ELOVO7, FJ47, FBXO7, GAK, GBA, GCDH, GCH1, GNAL, GNE, GRN, HPCA, KCTD17, KMT2B, LPIN1, LPIN2, LPIN3, LRRK2, MAPT, MCCC1, MCOLN1, NPC1, PANK2, PARK7, PDE8B, PDGFB PIN, PDGFR, PDGFR PLA2G, POLG, PRRKN, PRRKA, PSEN1, PSEN2, RAB12, RAB39B, SGCE excepto exón NM_001099401 exón 10, SLC19A3, SLC20A2, SLC30A10, SLC39A14, SLC6A3, SNCA, SNCB, SYN-1, SYNJ1, TA, TH1 TOR1A, VAC14, VPS13C (hotspot exones 11, 3, 4, 61 y 9), VPS35, XPR1 and agreed to participate in the study.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2024-07-01 (Estimated); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Change in non motor symptoms scale from baseline to 2 years | 2 years
  To determine the non motor symptoms profile and its evolution through non motor symptoms scale in glucocerebrosidase mutated Parkinson's disease in comparison with those without mutations. 30 items with total scores from 0 to 360, higher scores meaning higher non motor symptoms burden.
Change in non motor symptoms scale from baseline to 6 months | 6 months
  To determine the non motor symptoms profile and its evolution through non motor symptoms scale in glucocerebrosidase mutated Parkinson's disease in comparison with those without mutations. 30 items with total scores from 0 to 360, higher scores meaning higher non motor symptoms burden.
Change in non motor symptoms scale from 6 months to 1 year | 6 months
  To determine the non motor symptoms profile and its evolution through non motor symptoms scale in glucocerebrosidase mutated Parkinson's disease in comparison with those without mutations. 30 items with total scores from 0 to 360, higher scores meaning higher non motor symptoms burden.
Change in non motor symptoms scale from 12 months to 18 months | 6 months
  To determine the non motor symptoms profile and its evolution through non motor symptoms scale in glucocerebrosidase mutated Parkinson's disease in comparison with those without mutations. 30 items with total scores from 0 to 360, higher scores meaning higher non motor symptoms burden.
Change in non motor symptoms scale from 18 months to 24 months | 6 months
  To determine the non motor symptoms profile and its evolution through non motor symptoms scale in glucocerebrosidase mutated Parkinson's disease in comparison with those without mutations. 30 items with total scores from 0 to 360, higher scores meaning higher non motor symptoms burden.

SECONDARY OUTCOMES:
Change in Montreal Cognitive Assessment scale from baseline to 2 years | 2 years
  To determine the cognitive profile of glucocerebrosidase mutated Parkinson's disease in comparison with those without mutations, by using Montreal Cognitive Assessment. Scores ranging from 0 to 30, with lower scores meaning higher cognitive decline.
Change in Montreal Cognitive Assessment scale from baseline to 6 months | 6 months
  To determine the cognitive profile of glucocerebrosidase mutated Parkinson's disease in comparison with those without mutations, by using Montreal Cognitive Assessment. Scores ranging from 0 to 30, with lower scores meaning higher cognitive decline.
Change in Montreal Cognitive Assessment scale from 6 months to 12 months | 6 months
  To determine the cognitive profile of glucocerebrosidase mutated Parkinson's disease in comparison with those without mutations, by using Montreal Cognitive Assessment. Scores ranging from 0 to 30, with lower scores meaning higher cognitive decline.
Change in Montreal Cognitive Assessment scale from12 months to 18 months | 6 months
  To determine the cognitive profile of glucocerebrosidase mutated Parkinson's disease in comparison with those without mutations, by using Montreal Cognitive Assessment. Scores ranging from 0 to 30, with lower scores meaning higher cognitive decline.
Change in Montreal Cognitive Assessment scale from18 months to 24 months | 6 months
  To determine the cognitive profile of glucocerebrosidase mutated Parkinson's disease in comparison with those without mutations, by using Montreal Cognitive Assessment. Scores ranging from 0 to 30, with lower scores meaning higher cognitive decline.
Change in Parkinson's disease cognitive rating scale from baseline to 24 months | 2 years
  To determine the cognitive profile of glucocerebrosidase mutated Parkinson's disease in comparison with those without mutations, by using Parkinson's disease cognitive rating scale, scores from 0 to 134 with lower scores meaning higher cognitive decline.
Change in Parkinson's disease cognitive rating scale from baseline to 6 months | 6 months
  To determine the cognitive profile of glucocerebrosidase mutated Parkinson's disease in comparison with those without mutations, by using Parkinson's disease cognitive rating scale, scores from 0 to 134 with lower scores meaning higher cognitive decline.
Change in Parkinson's disease cognitive rating scale from 6 months to 12 months | 6 months
  To determine the cognitive profile of glucocerebrosidase mutated Parkinson's disease in comparison with those without mutations, by using Parkinson's disease cognitive rating scale, scores from 0 to 134 with lower scores meaning higher cognitive decline.
Change in Parkinson's disease cognitive rating scale from 12 months to 18 months | 6 months
  To determine the cognitive profile of glucocerebrosidase mutated Parkinson's disease in comparison with those without mutations, by using Parkinson's disease cognitive rating scale, scores from 0 to 134 with lower scores meaning higher cognitive decline.
Change in Parkinson's disease cognitive rating scale from 18 months to 24 months | 6 months
  To determine the cognitive profile of glucocerebrosidase mutated Parkinson's disease in comparison with those without mutations, by using Parkinson's disease cognitive rating scale, scores from 0 to 134 with lower scores meaning higher cognitive decline.
Change in Line Orientation Judgement scale from baseline to 24 months | 2 years
  To determine the cognitive profile of glucocerebrosidase mutated Parkinson's disease in comparison with those without mutations, by using Line Orientation Judgement, scores from 0 to 30 with lower punctuation meaning higher right hemisphere disfunction.
Change in Line Orientation Judgement scale from baseline to 6 months | 6 months
  To determine the cognitive profile of glucocerebrosidase mutated Parkinson's disease in comparison with those without mutations, by using Line Orientation Judgement, scores from 0 to 30 with lower punctuation meaning higher right hemisphere disfunction.
Change in Line Orientation Judgement scale from 6 months to 12 months | 6 months
  To determine the cognitive profile of glucocerebrosidase mutated Parkinson's disease in comparison with those without mutations, by using Line Orientation Judgement, scores from 0 to 30 with lower punctuation meaning higher right hemisphere disfunction.
Change in Line Orientation Judgement scale from 12 months to 18 months | 6 months
  To determine the cognitive profile of glucocerebrosidase mutated Parkinson's disease in comparison with those without mutations, by using Line Orientation Judgement, scores from 0 to 30 with lower punctuation meaning higher right hemisphere disfunction.
Change in Line Orientation Judgement scale from 18 months to 24 months | 6 months
  To determine the cognitive profile of glucocerebrosidase mutated Parkinson's disease in comparison with those without mutations, by using Line Orientation Judgement, scores from 0 to 30 with lower punctuation meaning higher right hemisphere disfunction.
Change in Rey figure from baseline to 24 months | 2 years
  To determine the cognitive profile of glucocerebrosidase mutated Parkinson's disease in comparison with those without mutations, by using Rey figure test, scoring from 0 to 72 points, meaning lower punctuations altered visuoperception and visual episodic memory.
Change in Rey figure from baseline to 6 months | 6 months
  To determine the cognitive profile of glucocerebrosidase mutated Parkinson's disease in comparison with those without mutations, by using Rey figure test, scoring from 0 to 72 points, meaning lower punctuations altered visuoperception and visual episodic memory.
Change in Rey figure from 6 months to 12 months | 6 months
  To determine the cognitive profile of glucocerebrosidase mutated Parkinson's disease in comparison with those without mutations, by using Rey figure test, scoring from 0 to 72 points, meaning lower punctuations altered visuoperception and visual episodic memory.
Change in Rey figure from 12 months to 18 months | 6 months
  To determine the cognitive profile of glucocerebrosidase mutated Parkinson's disease in comparison with those without mutations, by using Rey figure test, scoring from 0 to 72 points, meaning lower punctuations altered visuoperception and visual episodic memory.
Change in Rey figure from 18 months to 24 months | 6 months
  To determine the cognitive profile of glucocerebrosidase mutated Parkinson's disease in comparison with those without mutations, by using Rey figure test, scoring from 0 to 72 points, meaning lower punctuations altered visuoperception and visual episodic memory.
Change in Weschler Memory test from baseline to 24 months | 2 years
  To determine the cognitive profile of glucocerebrosidase mutated Parkinson's disease in comparison with those without mutations, by using Weschler Memory test, scoring in relation to age with percentiles from 0 to 100, lower percentile meaning a greater memory disturbance.
Change in Weschler Memory test from baseline to 6 months | 6 months
  To determine the cognitive profile of glucocerebrosidase mutated Parkinson's disease in comparison with those without mutations, by using Weschler Memory test, scoring in relation to age with percentiles from 0 to 100, lower percentile meaning a greater memory disturbance.
Change in Weschler Memory test from 6 months to 12 months | 6 months
  To determine the cognitive profile of glucocerebrosidase mutated Parkinson's disease in comparison with those without mutations, by using Weschler Memory test, scoring in relation to age with percentiles from 0 to 100, lower percentile meaning a greater memory disturbance.
Change in Weschler Memory test from 12 months to 18 months | 6 months
  To determine the cognitive profile of glucocerebrosidase mutated Parkinson's disease in comparison with those without mutations, by using Weschler Memory test, scoring in relation to age with percentiles from 0 to 100, lower percentile meaning a greater memory disturbance.
Change in Weschler Memory test from 18 months to 24 months | 6 months
  To determine the cognitive profile of glucocerebrosidase mutated Parkinson's disease in comparison with those without mutations, by using Weschler Memory test, scoring in relation to age with percentiles from 0 to 100, lower percentile meaning a greater memory disturbance.
Change in Stroop test from baseline to 24 months | 2 years
  To determine the cognitive profile of glucocerebrosidase mutated Parkinson's disease in comparison with those without mutations, by using Stroop test with T-scores from 0 to 100, higher scores reflecting better performance and less interference on reading ability.
Change in Stroop test from baseline to 6 months | 6 months
  To determine the cognitive profile of glucocerebrosidase mutated Parkinson's disease in comparison with those without mutations, by using Stroop test with T-scores from 0 to 100, higher scores reflecting better performance and less interference on reading ability.
Change in Stroop test from 6 months to 12 months | 6 months
  To determine the cognitive profile of glucocerebrosidase mutated Parkinson's disease in comparison with those without mutations, by using Stroop test with T-scores from 0 to 100, higher scores reflecting better performance and less interference on reading ability.
Change in Stroop test from 12 months to 18 months | 6 months
  To determine the cognitive profile of glucocerebrosidase mutated Parkinson's disease in comparison with those without mutations, by using Stroop test with T-scores from 0 to 100, higher scores reflecting better performance and less interference on reading ability.
Change in Stroop test from 18 months to 24 months | 6 months
  To determine the cognitive profile of glucocerebrosidase mutated Parkinson's disease in comparison with those without mutations, by using Stroop test with T-scores from 0 to 100, higher scores reflecting better performance and less interference on reading ability.
Change in Trail Making Test A from baseline to 24 months | 2 years
  To determine the cognitive profile of glucocerebrosidase mutated Parkinson's disease in comparison with those without mutations, by using Trail Making Test A, with scores ranging from 0 to 100 seconds, lower scores meaning better performance.
Change in Trail Making Test B from baseline to 24 months | 2 years
  To determine the cognitive profile of glucocerebrosidase mutated Parkinson's disease in comparison with those without mutations, by using Trail Making Test B, with scores ranging from 0 to 300 seconds, lower scores meaning better performance.
Change in Trail Making Test A from baseline to 6 months | 6 months
  To determine the cognitive profile of glucocerebrosidase mutated Parkinson's disease in comparison with those without mutations, by using Trail Making Test A, with scores ranging from 0 to 100 seconds, lower scores meaning better performance.
Change in Trail Making Test B from baseline to 6 months | 6 months
  To determine the cognitive profile of glucocerebrosidase mutated Parkinson's disease in comparison with those without mutations, by using Trail Making Test A, with scores ranging from 0 to 100 seconds, lower scores meaning better performance.
Change in Trail Making Test A from 6 months to 12 months | 6 months
  To determine the cognitive profile of glucocerebrosidase mutated Parkinson's disease in comparison with those without mutations, by using Trail Making Test B, with scores ranging from 0 to 300 seconds, lower scores meaning better performance.
Change in Trail Making Test B from 6 months to 12 months | 6 months
  To determine the cognitive profile of glucocerebrosidase mutated Parkinson's disease in comparison with those without mutations, by using Trail Making Test B, with scores ranging from 0 to 300 seconds, lower scores meaning better performance.
Change in Trail Making Test A from 12 months to 18 months | 6 months
  To determine the cognitive profile of glucocerebrosidase mutated Parkinson's disease in comparison with those without mutations, by using Trail Making Test A, with scores ranging from 0 to 100 seconds, lower scores meaning better performance.
Change in Trail Making Test B from 12 months to 18 months | 6 months
  To determine the cognitive profile of glucocerebrosidase mutated Parkinson's disease in comparison with those without mutations, by using Trail Making Test B, with scores ranging from 0 to 300 seconds, lower scores meaning better performance.
Change in Trail Making Test A from 18 months to 24 months | 6 months
  To determine the cognitive profile of glucocerebrosidase mutated Parkinson's disease in comparison with those without mutations, by using Trail Making Test A, with scores ranging from 0 to 100 seconds, lower scores meaning better performance.
Change in Trail Making Test B from 18 months to 24 months | 6 months
  To determine the cognitive profile of glucocerebrosidase mutated Parkinson's disease in comparison with those without mutations, by using Trail Making Test B, with scores ranging from 0 to 300 seconds, lower scores meaning better performance.
Change in Questionnaire for impulsive-compulsive disorders in Parkinson's disease (QUIP-RS) from baseline to 2 years | 2 years
  To determine impulse control disorder in glucocerebrosidase mutated Parkinson's disease in comparison with those without mutations, by using the Questionnaire for impulsive-compulsive disorders, scoring from 0 to 16 with lower scores meaning less impulsive-compulsive symptoms.
Change in Questionnaire for impulsive-compulsive disorders in Parkinson's disease (QUIP-RS) from baseline to 6 months | 6 months
  To determine impulse control disorder in glucocerebrosidase mutated Parkinson's disease in comparison with those without mutations, by using the Questionnaire for impulsive-compulsive disorders, scoring from 0 to 16 with lower scores meaning less impulsive-compulsive symptoms.
Change in Questionnaire for impulsive-compulsive disorders in Parkinson's disease (QUIP-RS) from 6 months to 12 months | 6 months
  To determine impulse control disorder in glucocerebrosidase mutated Parkinson's disease in comparison with those without mutations, by using the Questionnaire for impulsive-compulsive disorders, scoring from 0 to 16 with lower scores meaning less impulsive-compulsive symptoms.
Change in Questionnaire for impulsive-compulsive disorders in Parkinson's disease (QUIP-RS) from 12 months to 18 months | 6 months
  To determine impulse control disorder in glucocerebrosidase mutated Parkinson's disease in comparison with those without mutations, by using the Questionnaire for impulsive-compulsive disorders, scoring from 0 to 16 with lower scores meaning less impulsive-compulsive symptoms.
Change in Questionnaire for impulsive-compulsive disorders in Parkinson's disease (QUIP-RS) from 18 months to 24 months | 6 months
  To determine impulse control disorder in glucocerebrosidase mutated Parkinson's disease in comparison with those without mutations, by using the Questionnaire for impulsive-compulsive disorders, scoring from 0 to 16 with lower scores meaning less impulsive-compulsive symptoms.
Change in Neuropsychiatric inventory from baseline to 2 years | 2 years
  To determine neuropsychiatric profile in glucocerebrosidase mutated Parkinson's disease in comparison with those without mutations, by using Neuropsychiatric inventory, scoring from 0 to 144 with higher scores meaning greater neuropsychiatric symptoms.
Change in Neuropsychiatric inventory from baseline to 6 months | 6 months
  To determine neuropsychiatric profile in glucocerebrosidase mutated Parkinson's disease in comparison with those without mutations, by using Neuropsychiatric inventory, scoring from 0 to 144 with higher scores meaning greater neuropsychiatric symptoms.
Change in Neuropsychiatric inventory from 6 months to 12 months | 6 months
  To determine neuropsychiatric profile in glucocerebrosidase mutated Parkinson's disease in comparison with those without mutations, by using Neuropsychiatric inventory, scoring from 0 to 144 with higher scores meaning greater neuropsychiatric symptoms.
Change in Neuropsychiatric inventory from 12 months to 18 months | 6 months
  To determine neuropsychiatric profile in glucocerebrosidase mutated Parkinson's disease in comparison with those without mutations, by using Neuropsychiatric inventory, scoring from 0 to 144 with higher scores meaning greater neuropsychiatric symptoms.
Change in Neuropsychiatric inventory from 18 months to 24 months | 6 months
  To determine neuropsychiatric profile in glucocerebrosidase mutated Parkinson's disease in comparison with those without mutations, by using Neuropsychiatric inventory, scoring from 0 to 144 with higher scores meaning greater neuropsychiatric symptoms.
Change in Apathy Evaluation Scale from baseline to 24 months | 2 years
  To determine changes in apathy in glucocerebrosidase mutated Parkinson's disease in comparison with those without mutations, by using Apathy Evaluation Scale. The total score ranges from 18 to 72, with higher scores indicating more apathy.
Change in Apathy Evaluation Scale from baseline to 6 months | 6 months
  To determine changes in apathy in glucocerebrosidase mutated Parkinson's disease in comparison with those without mutations, by using Apathy Evaluation Scale. The total score ranges from 18 to 72, with higher scores indicating more apathy.
Change in Apathy Evaluation Scale from 6 months to 12 months | 6 months
  To determine changes in apathy in glucocerebrosidase mutated Parkinson's disease in comparison with those without mutations, by using Apathy Evaluation Scale. The total score ranges from 18 to 72, with higher scores indicating more apathy.
Change in Apathy Evaluation Scale from 12 months to 18 months | 6 months
  To determine changes in apathy in glucocerebrosidase mutated Parkinson's disease in comparison with those without mutations, by using Apathy Evaluation Scale. The total score ranges from 18 to 72, with higher scores indicating more apathy.
Change in Apathy Evaluation Scale from 18 months to 24 months | 6 months
  To determine changes in apathy in glucocerebrosidase mutated Parkinson's disease in comparison with those without mutations, by using Apathy Evaluation Scale. The total score ranges from 18 to 72, with higher scores indicating more apathy.
Change in Beck Depression Inventory from baseline to 24 months | 2 years
  To determine changes in depression in glucocerebrosidase mutated Parkinson's disease in comparison with those without mutations, by using Beck Depression Inventory with scores from 0 to 63, with higher scores meaning more depressive symptoms.
Change in Beck Depression Inventory from baseline to 6 months | 6 months
  To determine changes in depression in glucocerebrosidase mutated Parkinson's disease in comparison with those without mutations, by using Beck Depression Inventory with scores from 0 to 63, with higher scores meaning more depressive symptoms.
Change in Beck Depression Inventory from 6 months to 12 months | 6 months
  To determine changes in depression in glucocerebrosidase mutated Parkinson's disease in comparison with those without mutations, by using Beck Depression Inventory with scores from 0 to 63, with higher scores meaning more depressive symptoms.
Change in Beck Depression Inventory from 12 months to 18 months | 6 months
  To determine changes in depression in glucocerebrosidase mutated Parkinson's disease in comparison with those without mutations, by using Beck Depression Inventory with scores from 0 to 63, with higher scores meaning more depressive symptoms.
Change in Beck Depression Inventory from 18 months to 24 months | 6 months
  To determine changes in depression in glucocerebrosidase mutated Parkinson's disease in comparison with those without mutations, by using Beck Depression Inventory with scores from 0 to 63, with higher scores meaning more depressive symptoms.
Change in Stai-trait Anxiety Inventory from baseline to 24 months | 2 years
  To determine changes in anxiety in glucocerebrosidase mutated Parkinson's disease in comparison with those without mutations, by using State-trait Anxiety Inventory, scoring from 20 to 80, with higher punctuations meaning higher anxiety symptoms.
Change in Stai-trait Anxiety Inventory from baseline to 6 months | 6 months
  To determine changes in anxiety in glucocerebrosidase mutated Parkinson's disease in comparison with those without mutations, by using State-trait Anxiety Inventory, scoring from 20 to 80, with higher punctuations meaning higher anxiety symptoms.
Change in Stai-trait Anxiety Inventory from 6 months to 12 months | 6 months
  To determine changes in anxiety in glucocerebrosidase mutated Parkinson's disease in comparison with those without mutations, by using State-trait Anxiety Inventory, scoring from 20 to 80, with higher punctuations meaning higher anxiety symptoms.
Change in Stai-trait Anxiety Inventory from 12 months to 18 months | 6 months
  To determine changes in anxiety in glucocerebrosidase mutated Parkinson's disease in comparison with those without mutations, by using State-trait Anxiety Inventory, scoring from 20 to 80, with higher punctuations meaning higher anxiety symptoms.
Change in Stai-trait Anxiety Inventory from 18 months to 24 months | 6 months
  To determine changes in anxiety in glucocerebrosidase mutated Parkinson's disease in comparison with those without mutations, by using State-trait Anxiety Inventory, scoring from 20 to 80, with higher punctuations meaning higher anxiety symptoms.
Change in Parkinson's disease sleep scale from baseline to 24 months | 2 years
  To determine the sleep profile of glucocerebrosidase mutated Parkinson's disease in comparison with those without mutations, by using Parkinson's disease sleep scale, with scores from 0 to 150, the highest meaning less sleep symptoms.
Change in Parkinson's disease sleep scale from baseline to 6 months | 6 months
  To determine the sleep profile of glucocerebrosidase mutated Parkinson's disease in comparison with those without mutations, by using Parkinson's disease sleep scale, with scores from 0 to 150, the highest meaning less sleep symptoms.
Change in Parkinson's disease sleep scale from 6 months to 12 months | 6 months
  To determine the sleep profile of glucocerebrosidase mutated Parkinson's disease in comparison with those without mutations, by using Parkinson's disease sleep scale, with scores from 0 to 150, the highest meaning less sleep symptoms.
Change in Parkinson's disease sleep scale from 12 months to 18 months | 6 months
  To determine the sleep profile of glucocerebrosidase mutated Parkinson's disease in comparison with those without mutations, by using Parkinson's disease sleep scale, with scores from 0 to 150, the highest meaning less sleep symptoms.
Change in Parkinson's disease sleep scale from 18 months to 24 months | 6 months
  To determine the sleep profile of glucocerebrosidase mutated Parkinson's disease in comparison with those without mutations, by using Parkinson's disease sleep scale, with scores from 0 to 150, the highest meaning less sleep symptoms.
Change in Rapid Eye Movement Sleep Behavior Disorder Screening Questionnaire from baseline to 24 months | 2 years
  To determine the presence and symptoms of Rapid Eye Movement Sleep Behaviour Disorder in glucocerebrosidase mutated Parkinson's disease in comparison with those without mutations, by using Rapid Eye Movement Sleep Screening Questionnaire, scoring from 0 to 13 with higher scores meaning more Rapid Eye Movement sleep problems.
Change in REM Sleep Behavior Disorder Screening Questionnaire from baseline to 6 months | 6 months
  To determine the presence and symptoms of Rapid Eye Movement Sleep Behaviour Disorder in glucocerebrosidase mutated Parkinson's disease in comparison with those without mutations, by using Rapid Eye Movement Sleep Screening Questionnaire, scoring from 0 to 13 with higher scores meaning more Rapid Eye Movement sleep problems.
Change in REM Sleep Behavior Disorder Screening Questionnaire from to 6 months to 12 months | 6 months
  To determine the presence and symptoms of Rapid Eye Movement Sleep Behaviour Disorder in glucocerebrosidase mutated Parkinson's disease in comparison with those without mutations, by using Rapid Eye Movement Sleep Screening Questionnaire, scoring from 0 to 13 with higher scores meaning more Rapid Eye Movement sleep problems.
Change in REM Sleep Behavior Disorder Screening Questionnaire from to 12 months to 18 months | 6 months
  To determine the presence and symptoms of Rapid Eye Movement Sleep Behaviour Disorder in glucocerebrosidase mutated Parkinson's disease in comparison with those without mutations, by using Rapid Eye Movement Sleep Screening Questionnaire, scoring from 0 to 13 with higher scores meaning more Rapid Eye Movement sleep problems.
Change in REM Sleep Behavior Disorder Screening Questionnaire from to 18 months to 24 months | 6 months
  To determine the presence and symptoms of Rapid Eye Movement Sleep Behaviour Disorder in glucocerebrosidase mutated Parkinson's disease in comparison with those without mutations, by using Rapid Eye Movement Sleep Screening Questionnaire, scoring from 0 to 13 with higher scores meaning more Rapid Eye Movement sleep problems.
Change in Epworth Sleepiness Scale from baseline to 24 months | 2 years
  To determine the presence and severity of somnolence in glucocerebrosidase mutated Parkinson's disease in comparison with those without mutations, by using Epworth Sleepiness Scale, scoring from 0 to 24, with higher scores meaning higher sleeppiness.
Change in Epworth Sleepiness Scale from baseline to 6 months | 6 months
  To determine the presence and severity of somnolence in glucocerebrosidase mutated Parkinson's disease in comparison with those without mutations, by using Epworth Sleepiness Scale, scoring from 0 to 24, with higher scores meaning higher sleeppiness.
Change in Epworth Sleepiness Scale from 6 months to 12 months | 6 months
  To determine the presence and severity of somnolence in glucocerebrosidase mutated Parkinson's disease in comparison with those without mutations, by using Epworth Sleepiness Scale, scoring from 0 to 24, with higher scores meaning higher sleeppiness.
Change in Epworth Sleepiness Scale from 12 months to 18 months | 6 months
  To determine the presence and severity of somnolence in glucocerebrosidase mutated Parkinson's disease in comparison with those without mutations, by using Epworth Sleepiness Scale, scoring from 0 to 24, with higher scores meaning higher sleeppiness.
Change in Epworth Sleepiness Scale from 18 months to 24 months | 6 months
  To determine the presence and severity of somnolence in glucocerebrosidase mutated Parkinson's disease in comparison with those without mutations, by using Epworth Sleepiness Scale, scoring from 0 to 24, with higher scores meaning higher sleeppiness.
Change in Restless Legs Syndrome Rating Scale from baseline to 24 months | 2 years
  To determine the presence and severity of restless leg syndrome in glucocerebrosidase mutated Parkinson's disease in comparison with those without mutations, by using Restless Legs Syndrome Rating Scale, scoring from 0 to 40 with higher scores meaning greater restless legs syndrome symptoms.
Change in Restless Legs Syndrome Rating Scale from baseline to 6 months | 6 months
  To determine the presence and severity of restless leg syndrome in glucocerebrosidase mutated Parkinson's disease in comparison with those without mutations, by using Restless Legs Syndrome Rating Scale, scoring from 0 to 40 with higher scores meaning greater restless legs syndrome symptoms.
Change in Restless Legs Syndrome Rating Scale from 6 months to 12 months | 6 months
  To determine the presence and severity of restless leg syndrome in glucocerebrosidase mutated Parkinson's disease in comparison with those without mutations, by using Restless Legs Syndrome Rating Scale, scoring from 0 to 40 with higher scores meaning greater restless legs syndrome symptoms.
Change in Restless Legs Syndrome Rating Scale from 12 months to 18 months | 6 months
  To determine the presence and severity of restless leg syndrome in glucocerebrosidase mutated Parkinson's disease in comparison with those without mutations, by using Restless Legs Syndrome Rating Scale, scoring from 0 to 40 with higher scores meaning greater restless legs syndrome symptoms.
Change in Restless Legs Syndrome Rating Scale from 18 months to 24 months | 6 months
  To determine the presence and severity of restless leg syndrome in glucocerebrosidase mutated Parkinson's disease in comparison with those without mutations, by using Restless Legs Syndrome Rating Scale, scoring from 0 to 40 with higher scores meaning greater restless legs syndrome symptoms.
Change in Berg balance scale from baseline to 24 months | 2 years
  To determine changes in balance in glucocerebrosidase mutated Parkinson's disease in comparison with those without mutations, by using Berg Balance scale with ranges from 0 to 56. The lower score, the more at risk you of losing balance.
Change in Berg balance scale from baseline to 6 months | 6 months
  To determine changes in balance in glucocerebrosidase mutated Parkinson's disease in comparison with those without mutations, by using Berg Balance scale with ranges from 0 to 56. The lower score, the more at risk you of losing balance.
Change in Berg balance scale from 6 months to 12 months | 6 months
  To determine changes in balance in glucocerebrosidase mutated Parkinson's disease in comparison with those without mutations, by using Berg Balance scale with ranges from 0 to 56. The lower score, the more at risk you of losing balance.
Change in Berg balance scale from 12 months to 18 months | 6 months
  To determine changes in balance in glucocerebrosidase mutated Parkinson's disease in comparison with those without mutations, by using Berg Balance scale with ranges from 0 to 56. The lower score, the more at risk you of losing balance.
Change in Berg balance scale from 18 months to 24 months | 6 months
  To determine changes in balance in glucocerebrosidase mutated Parkinson's disease in comparison with those without mutations, by using Berg Balance scale with ranges from 0 to 56. The lower score, the more at risk you of losing balance.
Change in limits of stability from baseline to 24 months | 2 years
  To determine changes in balance in glucocerebrosidase mutated Parkinson's disease in comparison with those without mutations, by using % of performance regarding normalized limits of stability for reference sample, with values between 0-100%
Change in limits of stability from baseline to 6 months | 6 months
  To determine changes in balance in glucocerebrosidase mutated Parkinson's disease in comparison with those without mutations, by using % of performance regarding normalized limits of stability for reference sample, with values between 0-100%
Change in limits of stability from 6 months to 12 months | 6 months
  TTo determine changes in balance in glucocerebrosidase mutated Parkinson's disease in comparison with those without mutations, by using % of performance regarding normalized limits of stability for reference sample, with values between 0-100%
Change in limits of stability from 12 months to 18 months | 6 months
  To determine changes in balance in glucocerebrosidase mutated Parkinson's disease in comparison with those without mutations, by using % of performance regarding normalized limits of stability for reference sample, with values between 0-100%
Change in limits of stability from 18 months to 24 months | 6 months
  To determine changes in balance in glucocerebrosidase mutated Parkinson's disease in comparison with those without mutations, by using % of performance regarding normalized limits of stability for reference sample, with values between 0-100%
Change in speed reaction test from baseline to 24 months | 2 years
  To determine changes in speed reaction in glucocerebrosidase mutated Parkinson's disease in comparison with those without mutations, by using speed reaction tests measuring the time until response in seconds, with scores from 0 with no maximum value.
Change in speed reaction test from baseline to 6 months | 6 months
  TTo determine changes in speed reaction in glucocerebrosidase mutated Parkinson's disease in comparison with those without mutations, by using speed reaction tests measuring the time until response in seconds, with scores from 0 with no maximum value.
Change in speed reaction test from 6 months to 12 months | 6 months
  To determine changes in speed reaction in glucocerebrosidase mutated Parkinson's disease in comparison with those without mutations, by using speed reaction tests measuring the time until response in seconds, with scores from 0 with no maximum value.
Change in speed reaction test from 12 months to 18 months | 6 months
  To determine changes in speed reaction in glucocerebrosidase mutated Parkinson's disease in comparison with those without mutations, by using speed reaction tests measuring the time until response in seconds, with scores from 0 with no maximum value.
Change in speed reaction test from 18 months to 24 months | 6 months
  To determine changes in speed reaction in glucocerebrosidase mutated Parkinson's disease in comparison with those without mutations, by using speed reaction tests measuring the time until response in seconds, with scores from 0 with no maximum value.
Change in Movement Disorder's Society- Unified Parkinson's Disease Rating Scale part II scale from baseline to 24 months | 2 years
  To determine the motor profile of glucocerebrosidase mutated Parkinson's disease in comparison with those without mutations by using Movement Disorder's Society- Unified Parkinson's Disease Rating Scale part II, scoring from 0 to 52, higher scores meaning a greater Parkinson's symptoms burden.
Change in Movement Disorder's Society- Unified Parkinson's Disease Rating Scale part II from baseline to 6 months | 6 months
  To determine the motor profile of glucocerebrosidase mutated Parkinson's disease in comparison with those without mutations by using Movement Disorder's Society- Unified Parkinson's Disease Rating Scale part II, scoring from 0 to 52, higher scores meaning a greater Parkinson's symptoms burden.
Change in Movement Disorder's Society- Unified Parkinson's Disease Rating Scale part II from 6 months to 12 months | 6 months
  To determine the motor profile of glucocerebrosidase mutated Parkinson's disease in comparison with those without mutations by using Movement Disorder's Society- Unified Parkinson's Disease Rating Scale part II, scoring from 0 to 52, higher scores meaning a greater Parkinson's symptoms burden.
Change in Movement Disorder's Society- Unified Parkinson's Disease Rating Scale part II from 12 months to 18 months | 6 months
  To determine the motor profile of glucocerebrosidase mutated Parkinson's disease in comparison with those without mutations by using Movement Disorder's Society- Unified Parkinson's Disease Rating Scale part II, scoring from 0 to 52, higher scores meaning a greater Parkinson's symptoms burden.
Change in Movement Disorder's Society- Unified Parkinson's Disease Rating Scale part II from 18 months to 24 months | 6 months
  To determine the motor profile of glucocerebrosidase mutated Parkinson's disease in comparison with those without mutations by using Movement Disorder's Society- Unified Parkinson's Disease Rating Scale part II, scoring from 0 to 52, higher scores meaning a greater Parkinson's symptoms burden.
Change in Movement Disorder's Society- Unified Parkinson's Disease Rating Scale part III scale from baseline to 24 months | 2 years
  To determine the motor profile of glucocerebrosidase mutated Parkinson's disease in comparison with those without mutations by using Movement Disorder's Society- Unified Parkinson's Disease Rating Scale part III, scoring from 0 to 132, higher scores meaning a greater Parkinson's symptoms burden.
Change in Movement Disorder's Society- Unified Parkinson's Disease Rating Scale part III scale from baseline to 6 months | 6 months
  To determine the motor profile of glucocerebrosidase mutated Parkinson's disease in comparison with those without mutations by using Movement Disorder's Society- Unified Parkinson's Disease Rating Scale part III, scoring from 0 to 132, higher scores meaning a greater Parkinson's symptoms burden.
Change in Movement Disorder's Society- Unified Parkinson's Disease Rating Scale part III scale from 6 months to 12 months | 6 months
  To determine the motor profile of glucocerebrosidase mutated Parkinson's disease in comparison with those without mutations by using Movement Disorder's Society- Unified Parkinson's Disease Rating Scale part III, scoring from 0 to 132, higher scores meaning a greater Parkinson's symptoms burden.
Change in Movement Disorder's Society- Unified Parkinson's Disease Rating Scale part III scale from 12 months to 18 months | 6 months
  To determine the motor profile of glucocerebrosidase mutated Parkinson's disease in comparison with those without mutations by using Movement Disorder's Society- Unified Parkinson's Disease Rating Scale part III, scoring from 0 to 132, higher scores meaning a greater Parkinson's symptoms burden.
Change in Movement Disorder's Society- Unified Parkinson's Disease Rating Scale part III scale from 18 months to 24 months | 6 months
  To determine the motor profile of glucocerebrosidase mutated Parkinson's disease in comparison with those without mutations by using Movement Disorder's Society- Unified Parkinson's Disease Rating Scale part III, scoring from 0 to 132, higher scores meaning a greater Parkinson's symptoms burden.
Change in Movement Disorder's Society- Unified Parkinson's Disease Rating Scale part IV scale from baseline to 24 months | 2 years
  To determine the motor profile of glucocerebrosidase mutated Parkinson's disease in comparison with those without mutations by using Movement Disorder's Society- Unified Parkinson's Disease Rating Scale part IV, scoring from 0 to 24, higher scores meaning a greater Parkinson's symptoms burden.
Change in Movement Disorder's Society- Unified Parkinson's Disease Rating Scale part IV scale from baseline to 6 months | 6 months
  To determine the motor profile of glucocerebrosidase mutated Parkinson's disease in comparison with those without mutations by using Movement Disorder's Society- Unified Parkinson's Disease Rating Scale part IV, scoring from 0 to 24, higher scores meaning a greater Parkinson's symptoms burden.
Change in Movement Disorder's Society- Unified Parkinson's Disease Rating Scale part IV scale from 6 months to 12 months | 6 months
  To determine the motor profile of glucocerebrosidase mutated Parkinson's disease in comparison with those without mutations by using Movement Disorder's Society- Unified Parkinson's Disease Rating Scale part IV, scoring from 0 to 24, higher scores meaning a greater Parkinson's symptoms burden.
Change in Movement Disorder's Society- Unified Parkinson's Disease Rating Scale pary IV scale from 12 months to 18 months | 6 months
  To determine the motor profile of glucocerebrosidase mutated Parkinson's disease in comparison with those without mutations by using Movement Disorder's Society- Unified Parkinson's Disease Rating Scale part IV, scoring from 0 to 24, higher scores meaning a greater Parkinson's symptoms burden.
Change in Movement Disorder's Society- Unified Parkinson's Disease Rating Scale part IV scale from 18 months to 24 months | 6 months
  To determine the motor profile of glucocerebrosidase mutated Parkinson's disease in comparison with those without mutations by using Movement Disorder's Society- Unified Parkinson's Disease Rating Scale part IV, scoring from 0 to 24, higher scores meaning a greater Parkinson's symptoms burden.
Change in Hoehn and Yahr scale from baseline to 24 months | 2 years
  To determine the motor profile of glucocerebrosidase mutated Parkinson's disease in comparison with those without mutations by using Hoehn and Yahr scale, scores from 1-5, with lower scores meaning a lower motor symptom burden.
Change in Hoehn and Yahr scale from baseline to 6 months | 6 months
  To determine the motor profile of glucocerebrosidase mutated Parkinson's disease in comparison with those without mutations by using Hoehn and Yahr scale, scores from 1-5, with lower scores meaning a lower motor symptom burden.
Change in Hoehn and Yahr scale from 6 months to 12 months | 6 months
  To determine the motor profile of glucocerebrosidase mutated Parkinson's disease in comparison with those without mutations by using Hoehn and Yahr scale, scores from 1-5, with lower scores meaning a lower motor symptom burden.
Change in Hoehn and Yahr scale from 12 months to 18 months | 6 months
  To determine the motor profile of glucocerebrosidase mutated Parkinson's disease in comparison with those without mutations by using Hoehn and Yahr scale, scores from 1-5, with lower scores meaning a lower motor symptom burden.
Change in Hoehn and Yahr scale from 18 months to 24 months | 6 months
  To determine the motor profile of glucocerebrosidase mutated Parkinson's disease in comparison with those without mutations by using Hoehn and Yahr scale, scores from 1-5, with lower scores meaning a lower motor symptom burden.
Change in Parkinson's disease Questionnaire-39 from baseline to 24 months | 2 years
  To determine the repercusion of Parkinson's disease in daily activies in glucocerebrosidase mutated Parkinson's disease in comparison with those without mutations by using Parkinson's disease Questionnaire-39, scores from 0 to 100 with higher scores meaning greater repercussion in daily activities.
Change in Parkinson's disease Questionnaire-39 from baseline to 6 months | 6 months
  To determine the repercusion of Parkinson's disease in daily activies in glucocerebrosidase mutated Parkinson's disease in comparison with those without mutations by using Parkinson's disease Questionnaire-39, scores from 0 to 100 with higher scores meaning greater repercussion in daily activities.
Change in Parkinson's disease Questionnaire-39 from 6 months to 12 months | 6 months
  To determine the repercusion of Parkinson's disease in daily activies in glucocerebrosidase mutated Parkinson's disease in comparison with those without mutations by using Parkinson's disease Questionnaire-39, scores from 0 to 100 with higher scores meaning greater repercussion in daily activities.
Change in Parkinson's disease Questionnaire-39 from 12 months to 18 months | 6 months
  To determine the repercusion of Parkinson's disease in daily activies in glucocerebrosidase mutated Parkinson's disease in comparison with those without mutations by using Parkinson's disease Questionnaire-39, scores from 0 to 100 with higher scores meaning greater repercussion in daily activities.
Change in Parkinson's disease Questionnaire-39 from 18 months to 24 months | 6 months
  To determine the repercusion of Parkinson's disease in daily activies in glucocerebrosidase mutated Parkinson's disease in comparison with those without mutations by using Parkinson's disease Questionnaire-39, scores from 0 to 100 with higher scores meaning greater repercussion in daily activities.
Change in number of Parkinson's disease treatments from baseline to 24 months | 2 years
  To determine the changes in number of Parkinsons disease drugs during the course of the disease in glucocerebrosidase mutated Parkinson's disease in comparison with those without mutations.
Change in number of Parkinson's disease treatments from baseline to 6 months | 6 months
  To determine the changes in number of Parkinsons disease drugs during the course of the disease in glucocerebrosidase mutated Parkinson's disease in comparison with those without mutations.
Change in number of Parkinson's disease treatments from 6 months to 12 months | 6 months
  To determine the changes in number of Parkinsons disease drugs during the course of the disease in glucocerebrosidase mutated Parkinson's disease in comparison with those without mutations.
Change in number of Parkinson's disease treatments from 12 to 18 months | 6 months
  To determine the changes in number of Parkinsons disease drugs during the course of the disease in glucocerebrosidase mutated Parkinson's disease in comparison with those without mutations.
Change in number of Parkinson's disease treatments from 18 to 24 months | 6 months
  To determine the changes in number of Parkinsons disease drugs during the course of the disease in glucocerebrosidase mutated Parkinson's disease in comparison with those without mutations.

CONTACTS AND LOCATIONS:
Overall Officials: Inés Muro, MD, Principal Investigator — Hospital Universitario La Princesa; Juan P Romero, PhD, Study Director — Universidad Francisco de Vitoria; Lydia López, MD, Study Chair — Hospital Universitario La Princesa
Locations (2):
- Spain (2):
  - Universidad Francisco de Vitoria, Pozuelo de Alarcón, Madrid
  - Hospital Universitario La Princesa, Madrid

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Sidransky E, Nalls MA, Aasly JO, Aharon-Peretz J, Annesi G, Barbosa ER, Bar-Shira A, Berg D, Bras J, Brice A, Chen CM, Clark LN, Condroyer C, De Marco EV, Durr A, Eblan MJ, Fahn S, Farrer MJ, Fung HC, Gan-Or Z, Gasser T, Gershoni-Baruch R, Giladi N, Griffith A, Gurevich T, Januario C, Kropp P, Lang AE, Lee-Chen GJ, Lesage S, Marder K, Mata IF, Mirelman A, Mitsui J, Mizuta I, Nicoletti G, Oliveira C, Ottman R, Orr-Urtreger A, Pereira LV, Quattrone A, Rogaeva E, Rolfs A, Rosenbaum H, Rozenberg R, Samii A, Samaddar T, Schulte C, Sharma M, Singleton A, Spitz M, Tan EK, Tayebi N, Toda T, Troiano AR, Tsuji S, Wittstock M, Wolfsberg TG, Wu YR, Zabetian CP, Zhao Y, Ziegler SG. Multicenter analysis of glucocerebrosidase mutations in Parkinson's disease. N Engl J Med. 2009 Oct 22;361(17):1651-61. doi: 10.1056/NEJMoa0901281. PMID 19846850
- [Result] Barkhuizen M, Anderson DG, Grobler AF. Advances in GBA-associated Parkinson's disease--Pathology, presentation and therapies. Neurochem Int. 2016 Feb;93:6-25. doi: 10.1016/j.neuint.2015.12.004. Epub 2015 Dec 30. PMID 26743617
- [Result] Brockmann K, Srulijes K, Pflederer S, Hauser AK, Schulte C, Maetzler W, Gasser T, Berg D. GBA-associated Parkinson's disease: reduced survival and more rapid progression in a prospective longitudinal study. Mov Disord. 2015 Mar;30(3):407-11. doi: 10.1002/mds.26071. Epub 2014 Dec 1. PMID 25448271
- [Result] Leocadi M, Canu E, Donzuso G, Stojkovic T, Basaia S, Kresojevic N, Stankovic I, Sarasso E, Piramide N, Tomic A, Markovic V, Petrovic I, Stefanova E, Kostic VS, Filippi M, Agosta F. Longitudinal clinical, cognitive, and neuroanatomical changes over 5 years in GBA-positive Parkinson's disease patients. J Neurol. 2022 Mar;269(3):1485-1500. doi: 10.1007/s00415-021-10713-4. Epub 2021 Jul 23. PMID 34297177
- [Result] Swan M, Doan N, Ortega RA, Barrett M, Nichols W, Ozelius L, Soto-Valencia J, Boschung S, Deik A, Sarva H, Cabassa J, Johannes B, Raymond D, Marder K, Giladi N, Miravite J, Severt W, Sachdev R, Shanker V, Bressman S, Saunders-Pullman R. Neuropsychiatric characteristics of GBA-associated Parkinson disease. J Neurol Sci. 2016 Nov 15;370:63-69. doi: 10.1016/j.jns.2016.08.059. Epub 2016 Aug 30. PMID 27772789
- [Result] Malek N, Weil RS, Bresner C, Lawton MA, Grosset KA, Tan M, Bajaj N, Barker RA, Burn DJ, Foltynie T, Hardy J, Wood NW, Ben-Shlomo Y, Williams NW, Grosset DG, Morris HR; PRoBaND clinical consortium. Features of GBA-associated Parkinson's disease at presentation in the UK Tracking Parkinson's study. J Neurol Neurosurg Psychiatry. 2018 Jul;89(7):702-709. doi: 10.1136/jnnp-2017-317348. Epub 2018 Jan 29. PMID 29378790
- [Result] Ren J, Zhou G, Wang Y, Zhang R, Guo Z, Zhou H, Zheng H, Sun Y, Ma C, Lu M, Liu W. Association of GBA genotype with motor and cognitive decline in Chinese Parkinson's disease patients. Front Aging Neurosci. 2023 Feb 10;15:1091919. doi: 10.3389/fnagi.2023.1091919. eCollection 2023. PMID 36845659